CLINICAL TRIAL: NCT05247593
Title: The Efficacy and Safety of Dayingpian in The Treatment of Bipolar Disorder
Brief Title: A Study of Dayingpian Treating Bipolar Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, LI, Huafang, Executive Director of MICT, Shanghai Mental Health Center
Other Study IDs: SHDY2021CR2110C
Record Dates: First submitted 2022-02-16; First posted 2022-02-21 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Bipolar Disorder
Keywords: Cohort study; Bipolar disorder; Traditional Chinese Medicine; Efficacy; Dayingpian
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dayingpian exposure group 1: The exposure of interest is Dayingpian. Patients in this group take Dayingpian combined with conventional mood stabilizers. The psychiatrist does not assign specific interventions to the study participants. The course of observation is 12 weeks.
  Interventions: Drug: Dayingpian; Drug: conventional mood stabilizers
- Non-exposure group: The non-exposure group is the patients who do not take Dayingpian. Patients in this group take conventional mood stabilizers. The psychiatrist does not assign specific interventions to the study participants. The course of observation is 12 weeks.
  Interventions: Drug: conventional mood stabilizers
- Dayingpian exposure group 2: The exposure of interest is Dayingpian. Patients in this group take Dayingpian as monotherapy for bipolar disorder. The psychiatrist does not assign specific interventions to the study participants. The course of observation is 12 weeks.
  Interventions: Drug: Dayingpian

INTERVENTIONS:
Drug: Dayingpian — The actual dosage of Dayingpian is adjusted according to the patient's condition. The recommended dosage of Dayingpian is 5-10 tablets each time, 2-3 times a day.
  Groups: Dayingpian exposure group 1; Dayingpian exposure group 2
Drug: conventional mood stabilizers — Patients in the group are treated with the standard level of conventional mood stabilizers provided by psychiatrists according to treatment guidelines for bipolar disorder.
  Groups: Dayingpian exposure group 1; Non-exposure group

SUMMARY:
The main purpose of this cohort study is to evaluate the efficiency and safety of Dayingpian to provide evidence-based medical evidence for the subsequent drug development.

DETAILED DESCRIPTION:
Dayingpian is a kind of formula in traditional Chinese medicine with the effect of promoting blood circulation and reducing blood stasis. It has been prescribed as an add-on in the treatment of mental disorders such as bipolar disorder. However, there is not yet much high-quality evidence of the clinical effectiveness of Dayingpian treatment. In this study, we conduct a prospective, real-world longitudinal cohort study at Shanghai Mental Health Center in China to investigate the efficacy and safety of Dayingpian for bipolar disorder patients. The observation period is 12 weeks and all participants are evaluated every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the International Classification of Diseases-10(ICD-10) criteria for Bipolar Disorder.
2. Outpatients or inpatients in Shanghai Mental Health Center.
3. Male or female subjects aged 14-65 years.
4. education of Junior high school or above.
5. The patient fully understands and signs the informed consent form.

Exclusion Criteria:

1. Apparent violent aggression/suicide within the last two weeks.
2. Other patients that the investigator believes should not be included in the study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients or inpatients with bipolar disorder in Shanghai Mental Health Center are screened to participate in this study.
Sampling Method: Probability Sample
Enrollment: 308 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in the Young Mania Rating Scale (YMRS) scores compared with baseline | 12 weeks
  To assess the mania symptoms of bipolar disorder patients after 12 weeks of treatment. Patients are assessed with the scale at baseline and week 4, 8, 12(the end of study).

SECONDARY OUTCOMES:
Response rate | 12 weeks
  Response is defined as a reduction of at least 50% of the YMRS score compared with baseline.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) scores compared with baseline | 12 weeks
  To assess the depression symptoms of bipolar disorder patients after 12 weeks of treatment. Patients are assessed with the scale at baseline and week 4, 8, 12(the end of study).
Change in total score of the Clinical Global Impression-Severity (CGI-S) scale | 12 weeks
  To assess the severity of bipolar disorder with the scale at baseline and week 4, 8, 12(the end of study).
Change in total score of the Clinical Global Impression-Improvement (CGI-I) scale | 12 weeks
  To assess the improvement of bipolar disorder with the scale at baseline and week 4, 8, 12(the end of study).
Change of Traditional Chinese Medicine(TCM) syndromes scale | 12 weeks
  To assess the Traditional Chinese Medicine syndromes of patients with the scale at baseline and week 4, 8, 12(the end of study).

OTHER OUTCOMES:
Incidence of adverse events | 12 weeks
  Number of participants with adverse events during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No